CLINICAL TRIAL: NCT05424302
Title: Effect of Peripheral Vestibular Pathology Location on the Ability of Home-based Virtual Reality to Improve Symptoms of Peripheral Vestibular Disorders
Brief Title: Effect of Peripheral Vestibular Disease Location on Outcomes Following Home-based Virtual Reality Vestibular Therapy
Acronym: VR-PVD-RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Desmond A Nunez, Head, Division of Otolaryngology - Head and Neck Surgery, The University of British Columbia; Staff Otolaryngologist, Vancouver Hospital & Health Sciences Centre, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VR PVD RCT
Record Dates: First submitted 2022-02-15; First posted 2022-06-21 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Peripheral Vestibular Disorder; Benign Paroxysmal Positional Vertigo; Meniere Disease; Vestibular Neuritis; Vestibular Neuronitis; Labyrinthitis; Herpes Zoster Oticus
Keywords: Virtual reality; Video games; Peripheral vestibular disorders; Benign paroxysmal positional vertigo; Meniere disease; Vestibular Neuritis; Vestibular Neuronitis; Labyrinthitis; Herpes Zoster Oticus
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo; Meniere Disease; Vestibular Neuronitis; Labyrinthitis; Herpes Zoster Oticus

STUDY DESIGN:
Intervention Model Description: Patients will be divided into two groups using a computer-generated randomization schedule. These groups will undergo 4 or 8 weeks of vestibular rehabilitation for patients diagnosed with unilateral vestibular hypofunction or bilateral vestibular hypofunction respectively (Hall et al. 2016). This involves once a week 40-45 minute in-person sessions with a registered physiotherapist and three 20 minute sessions a day of at-home independent exercises (Hall et al. 2016). Standard vestibular rehabilitation involves a combination of exercises to promote gaze stability, to habituate symptoms, balance and gait training, and aerobic exercise (Hall et al. 2016). The virtual reality (VR) group will undergo an additional VR vestibular rehabilitation protocol. This will require them to utilize a head-mounted display device to play a video game projected on an android or apple device in a VR headset for 20 minutes daily until vestibular rehabilitation is complete (Micarelli et al. 2017, 2019).
Who Masked: Care Provider
Masking Description: The care provider(s) being masked to interventions assigned to participants in this clinical trial are the physiotherapists providing standard vestibular rehabilitation sessions to study participants. No other parties will be masked in this clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (Experimental): Patients have baseline data collected two weeks pre-intervention by assessing patient symptomatology using the dizziness handicap inventory, activities specific balance confidence questionnaires and a simulator sickness questionnaire remotely. Next, an interview will be conducted to collect information including age, sex, ethnicity, physical activity level and VR experience. Lastly, VR headset will be mailed to patients home address. A date for VR device tutorial will be discussed during this interview. Next patients will undergo 4 or 8 weeks of vestibular rehabilitation if diagnosed with unilateral or bilateral vestibular hypofunction respectively. This involves weekly 40-45 minute in-person sessions with a physiotherapist and three 20 minute sessions a day of at-home independent exercises. In addition, they will undergo an at home VR vestibular rehabilitation protocol that involves playing a video game projected on an android or apple device in a VR headset for 20 minutes daily.
  Interventions: Behavioral: Standard Vestibular Rehabilitation with Adjunct At Home Virtual Reality Vestibular Rehabilitation
- Control Group (Active Comparator): Patients have baseline data collected two weeks pre-intervention by assessing patient symptomatology using the dizziness handicap inventory, activities specific balance confidence questionnaires and a simulator sickness questionnaire remotely. Next, an interview will be conducted to collect information including age, sex, ethnicity, physical activity level and VR experience. Next patients will undergo 4 or 8 weeks of vestibular rehabilitation if diagnosed with unilateral or bilateral vestibular hypofunction respectively. This involves weekly 40-45 minute in-person sessions with a physiotherapist and three 20 minute sessions a day of at-home independent exercises. In addition, they will undergo an at-home regime that consists of auditory stimulation while wearing a VR headset for 20 minutes daily.
  Interventions: Behavioral: Standard Vestibular Rehabilitation with Adjunct Auditory Intervention

INTERVENTIONS:
Behavioral: Standard Vestibular Rehabilitation with Adjunct At Home Virtual Reality Vestibular Rehabilitation — The virtual reality intervention will involve standard vestibular rehabilitation as described above and adjunct at home virtual reality video game. This video game will be projected on an android or apple device accommodated into a VR headset for 20 minutes daily until the vestibular rehabilitation is complete. This video will be congruent to current vestibular rehabilitation program exercises. Point-of-view games compatible with both Android and iOS devices will be evaluated by professionals to determine the game that is most representative of current evidence based exercises.
  Arms: Virtual Reality Group
Behavioral: Standard Vestibular Rehabilitation with Adjunct Auditory Intervention — The control intervention will involve standard vestibular rehabilitation as described above and adjunct audio intervention while wearing the VR headset for 20 minutes daily until the vestibular rehabilitation is complete.
  Arms: Control Group

SUMMARY:
This parallel-group randomized controlled trial aims to determine if the location of the lesion(s) in the vestibular system (unilateral versus bilateral, lateral semi-circular canal versus otolith) impacts the effectiveness of adjunct take-home head-mounted display (HMD) virtual reality (VR) therapy in improving patient symptomatology. Fifty patients meeting inclusion criteria will be recruited from the principal investigator's neurotology clinic. Baseline symptomatology questionnaires will be completed, followed by random allocation to virtual reality and control groups. Vestibular rehabilitation and virtual reality protocols will be adhered to for 4 to 8 weeks, followed by symptomatology questionnaires. Data analysis will be conducted to answer the study's objectives.

DETAILED DESCRIPTION:
Purpose:

To determine if the location of the peripheral vestibular lesion(s) impacts the efficacy of adjunct at-home head-mounted display virtual reality therapy to improve patient symptomatology 0-3 months after the intervention. Also to determine the adverse effects caused by at-home head-mounted display virtual reality therapy.

Justification:

Home-based head-mounted display virtual reality video game exercises utilize a virtual environment to encourage wearers to complete head movements that mimic vestibular rehabilitation exercises. This virtual reality intervention could act as a valuable adjunct to standard virtual reality therapy. However, current literature lacks information on how the location of peripheral vestibular pathology impacts the efficacy of HBVR vestibular rehabilitation. Adding this information to the field could further personalize vestibular rehabilitation to the patient. Our research study personnel, specialist clinic, and access to vestibular investigations positions us well to undertake this work.

Research Design:

This is a parallel-group randomized controlled trial involving multiple clinical visits (the exact amount depends on diagnosis).

Statistical Analysis:

A sample size of 40 (20 per group) was determined to be sufficient for this study based on previous literature and the desired power that we hope to achieve. A meta-analysis completed by the research team, which is currently being considered for publication, indicated that the mean of the standardized mean DHI differences in current randomized controlled trials on VR in vestibular rehabilitation is -1.13. One article from this meta-analysis with a similar methodology to this RCT had a standardized mean ABC difference of 1.0. Additionally, well-designed randomized controlled trials set their type II error rate for 0.20 or 0.10 which results in a power of 80 or 90 percent. Inputting these standardized mean differences and 90% power values into the nomograph published by Altman 1982, yields a maximum sample size of 30 for DHI and 40 for ABC. Adopting the larger sample size and making an allowance for an acceptable attrition rate of 20%, it is proposed to recruit 50 patients in order to achieve a final sample size of 40 and thus a power of 90% for DHI and ABC data.

Mean and standard deviations will be calculated for each group's DHI and ABC scores 2 weeks before and after the intervention. Mean and standard deviations for patient SSQ scores will be calculated for each week of the protocol. An unpaired two-sample Wilcoxon test and a paired two-samples Wilcoxon test will be used to determine how significant the between (control vs. experimental) and in group (pre vs. post-treatment) differences are respectively. Subgroup analyses will be conducted on three subgroups of patients within each control and experimental group. These subgroups will be based on lesion location: lateral semicircular canal (Group A), utricle (Group B), and saccule (Group C). Matching subgroups from control and experimental groups will also be analyzed using unpaired two-samples Wilcoxon test and a paired two-samples Wilcoxon test to determine how significant the between (control vs. experimental) and in-group (pre vs. post-treatment) differences are respectively. Statistical significance cut-off (α) will be set at a p-value of 0.05.

Project Flow:

The patient will be contacted by phone or UBC Zoom conference call two weeks before the intervention begins to attain baseline data. This will involve assessing patient symptomatology by completing the dizziness handicap inventory (DHI) and activities-specific balance confidence (ABC) questionnaires remotely. Next, an interview will be conducted on this call to collect additional patient information including age, sex, ethnicity, physical activity level and virtual reality experience. Lastly, the VR headset will be mailed to the patient's home address using insured FedEx shipping. A date (before intervention start) for a VR device tutorial will be discussed at this visit.

Next, patients will be divided into two groups using a computer-generated randomization schedule. These groups will both undergo standard vestibular rehabilitation administered by a registered physiotherapist. This is considered standard of care and requires 4 to 8 weeks of vestibular rehabilitation for unilateral vestibular hypofunction (UVH) and bilateral vestibular hypofunction (BVH) respectively. This entails once a week 40 to 45-minute in-person sessions with a registered physiotherapist and 3 sessions a day of at-home exercises. The in-person sessions involve a combination of 4 different exercises: (1) exercises to promote gaze stability, (2) exercises to habituate symptoms, (3) balance and gait training, and (4) aerobic exercise. Gaze stability exercises that promote adaptation and substitution are both performed. Adaptation gaze stability exercises involve head movement while maintaining focus on a stationary or moving target. Substitution gaze stability exercises could include eye-head exercises where you conduct a large eye movement to a target before moving your head to face the target. Habituation exercises are conducted to expose the patient to dizziness-provoking stimuli in order to reduce symptoms to these stimuli over time. This could involve the use of optokinetic stimuli or virtual reality environments. Balance and gait training exercises are used to facilitate the use of visual and/or somatosensory inputs to substitute for lost vestibular function. Balance exercises involve balancing whilst experiencing altered visual input (ex. eyes closed) and/or somatosensory input (ex. foam or moving surface). Lastly, aerobic exercise, such as a stationary bicycle, is used for general conditioning because patients with vestibular hypofunction tend to limit physical activity to avoid symptom provocation. The registered physiotherapist providing this therapy will be blinded to patient group allocation. Patients will also complete 3 sessions a day of at-home adaptation, substitution, habituation, and balance exercises for a total of at least 20 minutes per day. The exact exercises will be similar to the in-person sessions however they will be truncated and adapted to the home setting.

Additionally, for 20 minutes per day for 4 (UVH) or 8 weeks (BVH) the virtual reality group will utilize a head-mounted display device to play a video game projected on an android or apple device accommodated into a VR headset. At-home exercises and VR usage will be recorded by patients using a study diary. Parameters recorded in the diary will include VR intervention usage (time of day, duration), physical activity (time of day, duration), and diet (breakfast, lunch and dinner contents and time of day). The patient will be instructed on how to size and use the VR headset during a tutorial scheduled after the initial assessment. A simulator sickness questionnaire (SSQ) will be completed every day after either the home exercise program (control group) or VR game intervention (experimental group). Two weeks after the intervention period patients will complete a subsequent remote assessment of symptomatology (DHI and ABC) and will return the VR headset through an insured FedEx shipment to Dr. Nunez's Neurotology clinic at the Gordon and Leslie Diamond Health Care Centre in Vancouver BC. VR headsets will be disinfected according to Vancouver coastal health protocols prior to providing the headset to subsequent patients. Additionally, both study groups will have submitted their study diary and SSQs to the research team via email or mail by this time.

Prior to completing the above interventions, the video game used must be congruent to current vestibular rehabilitation program exercises taught by a Canadian university physiotherapy program. The exact video game has not yet been chosen, however, point-of-view racing games compatible with both Android and iOS devices will be evaluated. This is due to Micarelli et al. 2017 and Micarelli et al. 2019 demonstrating the symptomatic benefits of this class of VR videogame. This evaluation will require a member of the research team to be filmed playing various point-of-view VR racing games. These videos will be sent to faculty and students at a Canadian University's Physiotherapy Program. After watching the videos, these individuals will complete a survey with 5-point Likert questions that ask for their opinion on if the video game effectively mimicked standard vestibular rehabilitation. The video game with the highest average score across all faculty members and students will be used by participants within the virtual reality intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with chronic (≥3 months) unilateral or bilateral peripheral vestibular disorders such as vestibular neuritis, labyrinthitis, Ramsay Hunt syndrome, ischemic lesion and trauma.
* Diagnosis made using caloric testing (≥25% reduced vestibular response) and either ocular vestibular evoked myogenic potential (oVEMP) or cervical vestibular evoked myogenic potential (cVEMP) testing.
* Participants prescribed vestibular rehabilitation
* Participants ≥18 years of age
* Access to an android or iOS smart phone

Exclusion Criteria:

* Pregnant participants
* Participant diagnosed with a central vestibular disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Dizziness Handicap Inventory (DHI) score | Change from baseline DHI score at 2 weeks post-intervention will be recorded for each patient.
  The Dizziness Handicap Inventory (DHI) score is a validated symptom index score created in 1990 that measures the functional, emotional and physical impacts of dizziness on the patient. This involves 25 questions which are answered as yes, sometimes or no. Yes response is 4 points, sometimes is 2 points and no is 0 points. The sum of these points are used to determine the severity of functional impairment. This severity is classified by the following ranges: mild 0-30, moderate 31-60 and severe 61-100.

SECONDARY OUTCOMES:
Activities-specific Balance Confidence (ABC) score | This ABC score will be calculated 2 weeks before intervention and 2 weeks after intervention.
  The ABC score is a validated measure of balance that includes 16 items which assesses balance confidence using a variety of activities with various difficulties. These 16 items are ranked from 0 (no confidence in completing task) to 100% (complete confidence in completing task).

OTHER OUTCOMES:
Simulator Sickness Questionnaire (SSQ) score | The SSQ will be completed at the baseline visit and every day of the home exercise program or virtual reality game intervention which can range from 28 days to 56 days depending on laterality of the peripheral vestibular disorder.
  The simulator sickness questionnaire is a validated tool for assessing simulator sickness which can help identify simulators that illicit significant side effects. Individuals are to rate the listed symptoms in the questionnaire using a four point scale: 0 (none), 1 (slight), 2 (moderate), 3 (severe). These individual symptom scores are multiplied by their listed weights and then summed for each Simulator Sickness Questionnaire (SSQ) section: Nausea (N), Oculomotor (O) and Disorientation (D). These total scores are inputted into a conversion formulas to get the individual N, O and D scores. Total score (TS) is calculated by summing all weighted totals and inputting them into a TS conversion formula above.

CONTACTS AND LOCATIONS:
Overall Officials: Desmond A Nunez, MD, MBA, Principal Investigator — Division of Otolaryngology, Department of Surgery, The University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
Results from this study will be analyzed and reported in the form of a publication in a scientific journal and or at neurotology conferences. These results may be published in an open-access journal, which means that there are no restrictions on who can access the data. Moreover, all deidentified individual participant raw data collected may be made available for other researchers to use in future projects. All published results and future studies that utilize our data will be sent to participants through email.
Supporting Information: Study Protocol
Time Frame: This time frame depends on the date of publication and the data registry guidelines.
Access Criteria: Data required by the data registry affiliated with the respective open access journal will be shared to enable publication of the manuscript.

REFERENCES:
- [Background] Micarelli A, Viziano A, Augimeri I, Micarelli D, Alessandrini M. Three-dimensional head-mounted gaming task procedure maximizes effects of vestibular rehabilitation in unilateral vestibular hypofunction: a randomized controlled pilot trial. Int J Rehabil Res. 2017 Dec;40(4):325-332. doi: 10.1097/MRR.0000000000000244. PMID 28723718
- [Background] Micarelli A, Viziano A, Micarelli B, Augimeri I, Alessandrini M. Vestibular rehabilitation in older adults with and without mild cognitive impairment: Effects of virtual reality using a head-mounted display. Arch Gerontol Geriatr. 2019 Jul-Aug;83:246-256. doi: 10.1016/j.archger.2019.05.008. Epub 2019 May 10. PMID 31102927
- [Background] Hall CD, Herdman SJ, Whitney SL, Cass SP, Clendaniel RA, Fife TD, Furman JM, Getchius TS, Goebel JA, Shepard NT, Woodhouse SN. Vestibular Rehabilitation for Peripheral Vestibular Hypofunction: An Evidence-Based Clinical Practice Guideline: FROM THE AMERICAN PHYSICAL THERAPY ASSOCIATION NEUROLOGY SECTION. J Neurol Phys Ther. 2016 Apr;40(2):124-55. doi: 10.1097/NPT.0000000000000120. PMID 26913496